CLINICAL TRIAL: NCT00175760
Title: Prospective Assessment of High Titre TTG to Diagnose Celiac Disease in Select Paediatric Patients.
Brief Title: Can a Very High Result From a Screening Test for Celiac Disease be Used to Diagnose Celiac Disease?
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Collin Barker, University of British Columbia
Other Study IDs: C04-0304
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Celiac Disease
Keywords: TTG; pediatric; comparison study
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Diagnosis of Celiac Disease — During GI endoscopy a minimum of 4 small intestinal biopsies will be taken from all subjects and controls.

SUMMARY:
This study is to see if a high response to the TTG screening test for celiac disease is as accurate as the current method of diagnosing celiac disease which entails a general anesthetic and upper endoscopy to obtain biopsies of the small intestine. If the screening blood test is highly accurate, then some patients that are being evaluated for celiac disease may not require an upper GI endoscopy and can be treated more quickly. If they respond to the therapy then they will be deemed to have celiac disease.

DETAILED DESCRIPTION:
All patients scheduled for upper GI endoscopy will be approached for recruitment into the study. A minimum of 4 small intestinal biopsies will be taken from all subjects and controls. All TTG specimens will be run through the hospital laboratory. Intermediate level TTG values 20-100 will be assessed separately and as part of the larger group. An optional part B of the study will assess the frequency of lactose intolerance in subjects prior to the start of a gluten free diet.

ELIGIBILITY:
Inclusion Criteria:

Inclusion-All patients planned to undergo upper GI endoscopy with biopsies.

Exclusion Criteria:

Exclusion-refusal to participate, not planning to have biopsies performed with the endoscopy.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Aged 2 months to 18 years with a planned upper GI endoscopy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-12; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Collin Barker, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada